CLINICAL TRIAL: NCT03901352
Title: An Asian, Multicenter, Randomized, Double-blind, Placebo-controlled, 14-week Study of Mirogabalin in Participants With Central Neuropathic Pain Followed by a 52-week, Open-label Extension
Brief Title: Study of Mirogabalin for Central Neuropathic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DS5565-A-J314; 194653 (Registry Identifier: JAPIC CTI)
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Central Neuropathic Pain
Keywords: Central neuropathic pain; Developmental phase III
MeSH Terms: interventions — mirogabalin

STUDY DESIGN:
Intervention Model Description: During the Double-blind Phase, participants will be randomized into parallel treatment arms.
  During the Open Extension Phase, all participants will be assigned to a single group.
Who Masked: Participant, Care Provider, Investigator
Masking Description: During the Double-blind Phase, masking will be triple (as shown above). During the Open Extension Phase, there will be no masking - the allocation is not applicable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirogabalin (Experimental): The patients with creatinine clearance (CLcr) ≥ 60 mL/min: Mirogabalin 20 mg or 30 mg, oral administration, Treatment period; 2-weeks titration and 12-weeks maintenance dose.
  The patients with creatinine clearance (CLcr) 30 to < 60 mL/min: Mirogabalin 10 mg or 15 mg, oral administration, Treatment period; 2-weeks titration and 12-weeks maintenance dose
  Interventions: Drug: Mirogabalin
- Placebo (Placebo Comparator): Placebo (14-weeks)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Matching placebo tablets for oral administration
  Other Names: Matching Placebo
  Arms: Placebo
Drug: Mirogabalin — Mirogabalin tablets for oral administration
  Other Names: DS-5565
  Arms: Mirogabalin

SUMMARY:
Investigate the efficacy and safety of mirogabalin in participants with central neuropathic pain in comparison to placebo

DETAILED DESCRIPTION:
[Double Blind Phase] The primary objective is to compare change in the Average Daily Pain Score (ADPS) from baseline to Week 14 in Asian participants with central neuropathic pain (central neuropathic pain after spinal cord injury) receiving mirogabalin versus placebo.

[Open Extension Phase] The objective is to assess the long-term safety and efficacy of mirogabalin in participants with central neuropathic pain (central neuropathic pain after spinal cord injury, central post stroke pain, and central neuropathic pain in Parkinson's disease).

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury (SCI) due to trauma
* American Spinal Injury Association impairment scale A, B, C, or D

Exclusion Criteria:

* Other severe pain at screening or randomization, unrelated to central neuropathic pain after SCI, that may confound the assessment of central neuropathic pain after SCI
* Neurologic disorders at screening or randomization, unrelated to central neuropathic pain after SCI, that may confound the assessment of central neuropathic pain after SCI
* Major psychiatric disorders within 1 year prior to screening

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2020-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Leader, Study Director — Daiichi Sankyo
Locations (118):
- Japan (101):
  - Chubu-Rosai Hospital, Aichi
  - Social Medical Corporation Daido Clinic, Aichi
  - Honmachi Clinic, Aichi
  - Nagoya City West Medical Center, Aichi
  - Toyota Kosei Hospital, Aichi
  - Nagoya Tokushukai General Hospital, Aichi
  - Kainan Hospital, Aichi
  - Hachinohe City Hospital, Aomori
  - Hirosaki University Hospital, Aomori
  - Chiba University Hospital, Chiba
  - Chiba Rehabilitation Center, Chiba
  - Funabashi Municipal Medical Center, Chiba
  - Kimitsu Chuo Hospital, Chiba
  - Ehime Prefectural Central Hospital, Ehime
  - University of Fukui Hospital, Fukui
  - Fukui-ken Saiseikai Hospital, Fukui
  - Shin Komonji Hospital, Fukuoka
  - Kyushu Rosai Hospital, Fukuoka
  - Steel Memorial Yawata Hospital, Fukuoka
  - Go Neurosurgical Clinic, Fukuoka
  - Japan Organization of Occupational Health and Safety Spinal Injuries Center, Fukuoka
  - Shin Yukuhashi Hospital, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Southern TOHOKU Medical Clinic, Fukushima
  - Japanese Red Cross Maebashi Hospital, Gunma
  - Goodlife Hospital, Hiroshima
  - Medical Corporation Suiseikai Suiseikai Kajikawa Hospital, Hiroshima
  - Hiroshima City Asa Citizens Hospital, Hiroshima
  - Hiroshima Prefectural Hospital, Hiroshima
  - Teine Keijinkai Hospital, Hokkaido
  - Hakodate Municipal Hospital, Hokkaido
  - Sapporo Medical University Hospital, Hokkaido
  - Nakamura Memorial Hospital, Hokkaido
  - Sapporo City General Hospital, Hokkaido
  - Japanese Red Cross Asahikawa Hospital, Hokkaido
  - Hokkaido Spinal Cord Injury Center, Hokkaido
  - Kobe City Medical Center General Hospital, Hyōgo
  - Japanese Red Cross Kobe Hospital, Hyōgo
  - Hyogo Social Welfare Corporation Hyogo Rehabilitation Center Central Hospital, Hyōgo
  - Japanese Red Cross Society Himeji Hospital, Hyōgo
  - University of Tsukuba Hospital, Ibaraki
  - Ibaraki Seinan Medical Center Hospital, Ibaraki
  - Ishikawa Prefectural Central Hospital, Ishikawa
  - Kagawa Prefectural Central Hospital, Kagawa
  - Shikoku Medical Center for Children and Adults, Kagawa
  - Japan Organization of Occupational Health and Safety(JOHAS), Yokohama Rosai Hospital, Kanagawa
  - Yokohama City Minato Red Cross Hospital, Kanagawa
  - Yokohama City University Hospital, Kanagawa
  - Kanagawa Rehabilitation Hospital, Kanagawa
  - Sagamihara Kyodo Hospital, Kanagawa
  - National Hospital Organaization Kumamoto Medical Center, Kumamoto
  - Kumamoto Kinoh Hospital, Kumamoto
  - Kumamoto Takumadai Rehabilitation Hospital, Kumamoto
  - Kumamoto Rehabilitation Hospital, Kumamoto
  - Uji-Tokushukai Medical Center, Kyoto
  - Mie University Hospital, Mie
  - Tohoku Rosai Hospital, Miyagi
  - National Hospital Organization Sendai Medical Center, Miyagi
  - Katta General Hospital, Miyagi
  - Junwakai Memorial Hospital, Miyazaki
  - University of Miyazaki Hospital, Miyazaki
  - Japan Red Cross Society Azumino Hospital, Nagano
  - Nagasaki University Hospital, Nagasaki
  - Nagasaki Rosai Hospital, Nagasaki
  - Nara Prefecture General Rehabilitation Center, Nara
  - Japanese Red Cross Society Nagaoka Red Cross Hospital, Niigata
  - Nagaoka Chuo General Hospital, Niigata
  - Niigata City General Hospital, Niigata
  - Niigata University Medical & Dental Hospital, Niigata
  - Iwate Rehabilitation Center, Numakunai
  - Okayama City General Medical Center Okayama City Hospital, Okayama
  - Kibikogen Rehabilitation Center For Employment Injuries, Okayama
  - Medical Corporation Tapic Okinawa Rehabilitation Center Hospital, Okinawa
  - Osaka General Medical Center, Osaka
  - Osaka University Hospital, Osaka
  - Aijinkai Rehabilitation Hospital, Osaka
  - Osaka Rosai Hospital, Osaka
  - Medical Corporation Keiaikai Nakamura Hospital, Ōita
  - Saga-ken Medical Centre KOSEIKAN, Saga
  - Hanyu General Hospital, Saitama
  - Otsu City Hospital, Shiga
  - Saiseikai Shiga Hospital, Shiga
  - Shimane University Hospital, Shimane
  - Shizuoka City Shimizu Hospital, Shizuoka
  - Fujieda Municipal General Hospital, Shizuoka
  - Hamamatsu University Hospital, Shizuoka
  - Japanese Red Cross Hamamatsu Hospital, Shizuoka
  - Kikugawa General Hospital, Shizuoka
  - Dokkyo Medical University Hospital, Tochigi
  - Jichi Medical University Hospital, Tochigi
  - Tokushima University Hospital, Tokushima
  - Makita General Hospital, Tokyo
  - Nihon University Itabashi Hospital, Tokyo
  - National Hospital Organaization Murayama Medical Center, Tokyo
  - Tottori University Hospital, Tottori
  - Toyama University Hospital Hospital, Toyama
  - Wakayama Medical University Hospital, Wakayama
  - Sanyudo Rehabilitation Center, Yamagata
  - Yamaguchi University Hospital, Yamaguchi
  - Yamaguchi Rosai Hospital, Yamaguchi
  - Yamanashi Prefectural Central Hospital, Yamanashi
- South Korea (13):
  - Daegu Fatima Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - CHA Bundang Medical Center, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - The Catholic University of Korea St. Vincent's Hospital, Gyeonggi-do
  - Ajou University Hospital, Gyeonggi-do
  - The Catholic University of Korea Incheon St. Mary's Hospital, Gyeonggi-do
  - Chonbuk National University Hospital, Jeollabuk-do
  - Pusan National University Hospital, Pusan
  - Pusan National University Yangsan Hospital, Pusan
  - Seoul Universtiy Hospital, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - Samsung Medical Center, Seoul
- Taiwan (4):
  - Hualien Tzu Chi Hospital, Hualien City
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: http://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Hosomi K, Katayama Y, Sakoda H, Kikumori K, Kuroha M, Ushida T. Usefulness of Mirogabalin in Central Neuropathic Pain After Stroke: Post Hoc Analysis of a Phase 3 Study by Stroke Type and Location. Pain Ther. 2024 Oct;13(5):1151-1171. doi: 10.1007/s40122-024-00616-3. Epub 2024 Jul 4. PMID 38963656
- [Derived] Ushida T, Katayama Y, Hiasa Y, Nishihara M, Tajima F, Katoh S, Tanaka H, Maeda T, Furusawa K, Kakehi Y, Kikumori K, Kuroha M. Long-Term Safety and Efficacy of Mirogabalin for Central Neuropathic Pain: A Multinational, Phase 3, 52-Week, Open-Label Study in Asia. Pain Ther. 2023 Aug;12(4):963-978. doi: 10.1007/s40122-023-00513-1. Epub 2023 Apr 28. PMID 37115464
- [Derived] Ushida T, Katayama Y, Hiasa Y, Nishihara M, Tajima F, Katoh S, Tanaka H, Maeda T, Furusawa K, Richardson M, Kakehi Y, Kikumori K, Kuroha M. Mirogabalin for Central Neuropathic Pain After Spinal Cord Injury: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study in Asia. Neurology. 2023 Mar 14;100(11):e1193-e1206. doi: 10.1212/WNL.0000000000201709. Epub 2022 Dec 14. PMID 36517235

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 300 participants who met all inclusion and no exclusion criteria were randomized to treatment at 118 study sites in Japan, South Korea, and Taiwan.
Pre-assignment Details: Participants being treated underwent a washout period ≥28 days. Mirogabalin starting dose and titration schedule were based on creatinine clearance per the Japanese drug insert. All mirogabalin patients who received any dose were assessed as 1 group for efficacy/safety as prespecified in the protocol.
Groups:
- Mirogabalin: Patients with creatinine clearance (CLcr) ≥ 60 mL/min were randomized to receive mirogabalin 20 mg or 30 mg by oral administration with a 2-weeks titration period and 12-weeks maintenance period.
  Patients with creatinine clearance (CLcr) 30 to < 60 mL/min were randomized to receive mirogabalin 10 mg or 15 mg by oral administration with a 2-weeks titration period and 12-weeks maintenance period.
- Placebo: Patients who received placebo for 14 weeks by oral administration.
Period: Double-blind Phase
Arm/Group | Mirogabalin | Placebo
Started | 150 | 150
Completed | 133 | 136
Not Completed | 17 | 14
Not completed — Adverse Event | 6 | 4
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 10 | 8
Period: Open-label Extension Phase
Arm/Group | Mirogabalin | Placebo
Started | 210 (Participants only received mirogabalin (low, medium, or high modal dose) in the open-label, long-term extension phase.) | 0 (No participants received placebo during the open-label, long-term extension phase.)
Completed | 170 | 0
Not Completed | 40 | 0
Not completed — Adverse Event | 24 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 14 | 0
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: Data were based on the modified Intent-to-Treat population (mITT). Mirogabalin starting dose and titration schedule were based on creatinine clearance per the Japanese drug insert. All mirogabalin patients who received any dose were assessed as 1 group for efficacy/safety as prespecified in the protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mirogabalin | Placebo | Total
Number analyzed (Participants) | 150 | 149 | 299
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 93 | 89 | 182
  >=65 years | 57 | 60 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (14.3) | 59.6 (14.0) | 58.5 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 24 | 43
  Male | 131 | 125 | 256
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 150 | 149 | 299
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 19 | 16 | 35
  Japan | 121 | 121 | 242
  Taiwan | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Weekly Average Daily Pain Score (ADPS) at Week 14 Following Administration With Mirogabalin or Placebo
Description: The pain scores on a scale of 0-10, where 0 = no pain and 10 = the worst possible pain. Negative changes in ADPS indicated an improvement in pain scores. The weekly ADPS is based on participants daily pain scores.
Time Frame: Baseline to Week 14 postdose
Population: Data were assessed in the mITT population. Mirogabalin starting dose and titration schedule were based on creatinine clearance per the Japanese drug insert. All mirogabalin patients who received any dose were assessed as 1 group for efficacy/safety as prespecified in the protocol.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Mirogabalin | Placebo
Number analyzed (Participants) | 150 | 149
units on a scale | -1.23 (0.132) | -0.52 (0.132)
Statistical Analysis 1: Comparison: Mirogabalin vs Placebo; Test type: Superiority; p = 0.0001, ANCOVA; Difference of LSM vs placebo = -0.71, 95% CI 2-sided [-1.08 to -0.34], Standard Error of Mean 0.187 — The multiple imputation (MI) was based on a "nonfuture dependence" model using the pattern mixture model (PMM) approach with shifting parameters under the missing not at random (MNAR0 mechanism for the missing weekly ADPS

2. Secondary Outcome: Number of Participants With ≥30% Reduction and ≥50% Reductions From Baseline in Average Daily Pain Score (ADPS)
Description: Responder rate (%) = 100 × (observed weekly ADPS - baseline weekly ADPS) / baseline weekly ADPS, where the baseline weekly ADPS was defined as the average of up to 7 available pain scores in the last 7 days at or before the randomization visit (Visit 2).
Time Frame: Baseline to Week 14 postdose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Mirogabalin | Placebo
Number analyzed (Participants) | 150 | 149
Participants
  ≥30% reduction from baseline at Week 14 | 46 | 28
  ≥50% reduction from baseline at Week 14 | 21 | 9

3. Secondary Outcome: Change From Baseline in Present Pain Intensity on the Short Form-McGill Pain Questionnaire at Week 14 Following Administration With Mirogabalin or Placebo
Description: Participants rated their present pain intensity on a scale of 0 (no pain) to 5 (most intense pain). Negative changes in present pain intensity indicated an improvement in pain intensity.
Time Frame: Baseline to Week 14 postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mirogabalin | Placebo
Number analyzed (Participants) | 150 | 149
units on a scale | -0.6 (0.92) | -0.3 (0.95)

4. Secondary Outcome: Patient Global Impression of Change at Week 14 Following Administration With Mirogabalin or Placebo
Description: At the end-of-treatment (Visit 7)/early termination visit, participants provided a self-assessment of their condition compared to the randomization visit (Visit 2) using the 7-point scale in the Patient Global Impression of Change (PGIC), where 1 = very much improved to 7 = very much worse. Here, the PGIC responder rates were categorized and defined as the percentage of participants who satisfied the following PGIC score criteria: Minimally improved or better (ie, score ≤3); Much improved or better (ie, score ≤2). Patient Global Impression of Change scores are used to determine categorical responder rates.
Time Frame: at Week 14 postdose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Mirogabalin | Placebo
Number analyzed (Participants) | 150 | 149
Participants
  Much improved or better (≤2) | 26 | 11
  Minimally improved or better (≤3) | 80 | 53

5. Secondary Outcome: Change From Baseline in the Weekly Average Daily Sleep Interference Score (ADSIS) Following Administration With Mirogabalin or Placebo
Description: The daily sleep interference diary consisted of an 11-point numerical rating scale (NRS) which was used to assess how pain had interfered with the participant's sleep during the past 24 hours. Participants recorded a sleep interference score in the patient diary once daily from the day after the screening visit (Visit 1) through the end-of-treatment (Visit 7)/early termination visit. Every morning upon awakening, prior to taking the study drug, each participant selected the number that best described his/her sleep interference experience during the past 24 hours on a scale of 0 = pain did not interfere with sleep to 10 = pain completely interfered with sleep. Negative values indicate an improvement in sleep interference. The weekly average daily sleep interference score (ADSIS) was based on the sleep interference scores from the patient diaries.
Time Frame: Baseline to Week 14 postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mirogabalin | Placebo
Number analyzed (Participants) | 150 | 149
units on a scale | -1.14 (1.705) | -0.35 (1.306)

6. Secondary Outcome: Change From Baseline in the Medical Outcomes Study Sleep Scale Scores Following Administration With Mirogabalin or Placebo
Description: The MOS sleep scale was based on questions about sleep quality during the past 4 weeks and consisted of 3 parts. Average time required to fall asleep, average hours of sleep per night, and ten questions based on sleep disturbance that were given a score of 1 (all the time) to 5 (none of the time). Based on the 12 questions, the following scales were calculated: sleep disturbance, snoring, awakening due to shortness of breath or headache, sleep adequacy, sleep somnolence, 9-item sleep item index, sleep quantity, and optimal sleep (not reported since it is a yes/no response). Each scale was given a score ranging from 1 (all the time) to 5 (none of the time), except for the 9-item sleep item index. Individual item scores of the 9-item sleep index were averaged and the total score ranged from 1 to 5. For all items reported, higher scores indicate an improvement in sleep disturbance.
Time Frame: Baseline to Week 14 postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mirogabalin | Placebo
Number analyzed (Participants) | 150 | 149
score on a scale
  Sleep disturbance | 4.23 (8.39) | 1.27 (7.15)
  Snoring | -1.12 (7.89) | 0.61 (7.73)
  Awakening due to shortness of breath or headache | 2.04 (12.64) | 0.71 (9.90)
  Sleep adequacy | 1.94 (9.87) | 0.81 (8.44)
  Sleep somnolence | -1.18 (10.04) | -0.05 (7.85)
  9-item sleep problems index | 2.70 (7.74) | 1.29 (6.15)
  Sleep quantity | 0.3 (1.46) | 0.1 (0.93)

7. Secondary Outcome: Change From Baseline in the Hospital Anxiety & Depression Scale Following Administration With Mirogabalin or Placebo
Description: The Hospital Anxiety and Depression (HADS) scale consisted of 7 items to score depression (4-point scale: 0 to 3; where a score of 3 indicates highest depression levels [worse outcome]) and 7 items to score anxiety (4-point scale: 0 to 3; where score of 3 indicates highest anxiety levels [worse outcome]). The depression and anxiety subscales were calculated by summing the corresponding scores for 7 items. Negative scores indicate an improvement in depression and anxiety.
Time Frame: Baseline to Week 14 postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mirogabalin | Placebo
Number analyzed (Participants) | 150 | 149
score on a scale
  Depression | -0.8 (3.18) | -0.7 (2.85)
  Anxiety | -1.0 (3.20) | -0.8 (2.85)

8. Secondary Outcome: Change From Baseline in the Neuropathic Pain Symptom Inventory Score Following Administration With Mirogabalin or Placebo
Description: The Neuropathic Pain Symptom Inventory assessment was comprised of 4 distinct dimensions of neuropathic pain: spontaneous pain, paroxysmal pain, evoked pain, and paresthesia/dysesthesia. Each dimension was scored on an 11-point scale from 0 (no pain) to 10 (the most intense pain imaginable) for reporting the mean intensity of each item of the dimension during the last 24 hours. The total score is the sum of each of the 4 dimensions of neuropathic pain and total score ranged from 0 to 40. Higher scores indicated worse outcome; negative values indicate an improvement.
Time Frame: Baseline to Week 14 postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mirogabalin | Placebo
Number analyzed (Participants) | 150 | 149
score on a scale
  Spontaneous pain | -4.2 (5.66) | -1.5 (6.17)
  Paroxysmal pain | -2.5 (4.40) | -0.9 (4.78)
  Evoked pain | -2.6 (5.80) | -1.0 (6.52)
  Paresthesia/dysesthesia | -2.7 (4.29) | -1.2 (3.67)
  Total score | -12.0 (15.47) | -4.5 (15.90)

9. Secondary Outcome: Change From Baseline in the EuroQoL 5 Dimensions 5 Levels Following Administration With Mirogabalin or Placebo
Description: The EuroQoL 5 Dimensions 5 Levels (EuroQoL-5D-5L) questionnaire yielded a 5-scale profile of the participant's self-assessed quality of life in each of the following dimensions: mobility (5-point scale), self-care (5-point scale), usual activities (5-point scale), pain/discomfort (5-point scale), and anxiety/depression (5-point scale). These profiles were combined into an overall health utilities index, and a visual analog scale (VAS) that measured the participants' perceptions of overall health. EQ-5D-5L index scores range from -0.59 (worst health state) to 1 (best possible health state). EQ VAS scores range from 0 (worse imaginable health or worst outcome) to 100 (best imaginable health or best outcome). Higher scores for index value and VAS indicate better outcome.
Time Frame: Baseline to Week 14 postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mirogabalin | Placebo
Number analyzed (Participants) | 150 | 149
score on a scale
  Index value | 0.0395 (0.136) | 0.0153 (0.134)
  Visual analog scale | 4.9 (21.76) | -1.8 (21.28)

10. Secondary Outcome: Change From Baseline in the Spinal Cord Independence Measure Scores Following Administration With Mirogabalin or Placebo
Description: The Spinal Cord Independence Measure (SCIM) score assessed the participants' activities of daily living (ADL). The SCIM instrument yielded a profile of the participant's ADL in the following categories: total SCIM score (0 to 100), self-care (scored 0 to 20; with higher scores indicating better self care), respiration and sphincter management (0 to 40; with higher scores indicating better management), and mobility (0 to 40; with higher scores indicating better mobility). Overall higher scores indicated better outcomes.
Time Frame: Baseline to Week 14 postdose
Population: Participants with available data were assessed in mITT population. Mirogabalin starting dose and titration schedule were based on creatinine clearance per the Japanese drug insert. All mirogabalin patients who received any dose were assessed as 1 group for efficacy/safety as prespecified in the protocol.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mirogabalin | Placebo
Number analyzed (Participants) | 149 | 149
score on a scale
  Self care | 0.3 (1.61) | 0 (1.59)
  Respiration and sphincter management | 0.7 (2.90) | 0 (3.21)
  Mobility | 0 (2.45) | 0 (1.68)
  Total score | 1.0 (4.71) | 0 (4.70)

11. Secondary Outcome: Number of Participants Who Performed At Level or Below Level for Allodynia Following Administration With Mirogabalin or Placebo
Description: Study investigators performed the test for allodynia (at level, below level) using a scale assessing the presence (at level) or absence (below level) of allodynia. Testing usually requires an external stimulation of non-painful quality.
Time Frame: Baseline to Week 14 postdose
Population: Participants with available data in mITT population were assessed. Mirogabalin starting dose and titration schedule were based on creatinine clearance per the Japanese drug insert. All mirogabalin patients who received any dose were assessed as 1 group for efficacy/safety as prespecified in the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Mirogabalin | Placebo
Number analyzed (Participants) | 49 | 50
Participants
  Below Level | 10 | 13
  At Level: number analyzed (Participants) | 29 | 34
  At Level | 5 | 6

12. Secondary Outcome: Change From Baseline in Present Pain Intensity on the Short Form-McGill Pain Questionnaire at Week 52 Following Administration With Mirogabalin During the Long-term Extension (LTE)
Description: Participants rated their present pain intensity on a visual analog scale of 0 (no pain) to 5 (most intense pain). Higher scores indicate worse outcome; negative changes in present pain intensity indicated an improvement in pain intensity.
Time Frame: Baseline to Week 52 postdose
Population: Data were assessed in the mITT population in the LTE phase. Mirogabalin starting dose and titration schedule were based on creatinine clearance per the Japanese drug insert. All mirogabalin patients who received any dose were assessed as 1 group for efficacy/safety as prespecified in the protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mirogabalin
Number analyzed (Participants) | 210
units on a scale | -9.6 (24.70)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline up to 52 weeks postdose.
Description: Mirogabalin starting dose and titration schedule were based on creatinine clearance per the Japanese drug insert. All mirogabalin patients who received any dose were assessed as 1 group for efficacy/safety as prespecified in the protocol.
Groups:
- Mirogabalin Open-Label Extension: Participants with creatinine clearance (CLcr) ≥60 mL/min who received 5 mg twice daily (BID) of mirogabalin in the first 2 weeks, followed by 10 mg BID in the second 2 weeks. From the fifth week on, if no safety concerns were raised, the dosage was increased to 15 mg BID. For the following weeks, the dosage could be either 10 mg BID or 15 mg BID, depending on the safety findings at each visit. During the last week of the treatment period, participants underwent tapering, receiving half of the daily dose received just before tapering.
  Participants with CLcr 30 to <60 mL/min received half of the dose of mirogabalin as participants with CLcr ≥60 mL/min during the treatment period.
Arm/Group | Mirogabalin | Placebo | Mirogabalin Open-Label Extension
All-Cause Mortality (participants affected / at risk) | 1/151 | 0/148 | 0/210
Serious Adverse Events (participants affected / at risk) | 9/151 | 7/148 | 28/210
Other Adverse Events (participants affected / at risk) | 112/151 | 34/148 | 178/210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mirogabalin (N=151) | Placebo (N=148) | Mirogabalin Open-Label Extension (N=210)
Cellulitis (Infections and infestations) | 2 | 0 | 2
Pneumonia (Infections and infestations) | 1 | 1 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Ranula (Gastrointestinal disorders) | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Cardiac death (General disorders) | 1 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Inflammation of wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 2
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 2
Breast cellulitis (Infections and infestations) | 0 | 0 | 1
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 1
Puncture site infection (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Diabetic retinopathy (Eye disorders) | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Neurogenic bladder (Renal and urinary disorders) | 0 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 1
Disuse syndrome (General disorders) | 0 | 0 | 1
Prolapse (General disorders) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cataract operation (Surgical and medical procedures) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mirogabalin (N=151) | Placebo (N=148) | Mirogabalin Open-Label Extension (N=210)
Nasopharyngitis (Infections and infestations) | 12 | 8 | 23
Somnolence (Nervous system disorders) | 45 | 8 | 35
Dizziness (Nervous system disorders) | 13 | 5 | 16
Constipation (Gastrointestinal disorders) | 9 | 2 | 13
Oedema peripheral (General disorders) | 9 | 2 | 26
Weight increased (Investigations) | 11 | 1 | 15
Urinary tract infection (Infections and infestations) | 5 | 5 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 11
Oedema (General disorders) | 5 | 0 | 24
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/52/NCT03901352/Prot_SAP_000.pdf